CLINICAL TRIAL: NCT00052390
Title: A Multi-Institutional, Open-Label, Phase II Study Of Doxorubicin And Bevacizumab (Anti-VEFG Monoclonal Antibody, NSC 704865) For Patients With Advanced Or Metastatic Soft-Tissue Sarcoma
Brief Title: Doxorubicin and Bevacizumab in Treating Patients With Locally Recurrent or Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258249; MSKCC-02041; NCI-2270
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2004-02

CONDITIONS: Sarcoma
Keywords: recurrent adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Bevacizumab; Doxorubicin

INTERVENTIONS:
Biological: bevacizumab
Drug: doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Bevacizumab may stop the growth of tumor cells by stopping blood flow to the tumor. Combining doxorubicin with bevacizumab may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining doxorubicin with bevacizumab in treating patients who have locally recurrent or metastatic soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate (partial and complete) in patients with locally recurrent or metastatic soft tissue sarcoma treated with doxorubicin and bevacizumab.
* Determine the tolerability of this regimen in these patients.
* Determine the toxicity profile of this regimen in these patients.
* Determine whether pre-treatment plasma vascular endothelial growth factor level or microvessel density of tumor samples from these patients predicts response to this regimen.

OUTLINE: This is a multicenter study.

Patients receive doxorubicin IV over 5-10 minutes followed by bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Patients with responding disease after reaching the maximum dose of doxorubicin may continue bevacizumab alone.

Patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 17-37 patients will be accrued for this study within 13.3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed soft tissue sarcoma

  * Locally recurrent or metastatic disease
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
* No prior or concurrent known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 80-100% OR
* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* No bleeding diathesis or coagulopathy

Hepatic

* Bilirubin no greater than 1.2 mg/dL
* AST and ALT no greater than 2.5 times upper limit of normal
* PT and aPTT normal

Renal

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min
* No proteinuria (must be less than 500 mg protein per 24 hours)

Cardiovascular

* Cardiac ejection fraction at least 50% by echocardiogram or MUGA
* No history of deep vein thrombosis
* No clinically significant cardiovascular disease
* No uncontrolled hypertension
* No myocardial infarction
* No unstable angina
* No New York Heart Association grade II-IV congestive heart failure
* No serious cardiac arrhythmia requiring medication
* No grade II or greater peripheral vascular disease within the past year

Pulmonary

* No history of pulmonary embolism

Other

* No symptomatic peripheral neuropathy grade 2 or greater
* No other neoplastic disease within the past 5 years except curatively treated basal cell skin cancer or carcinoma in situ of the cervix
* No prior allergic reactions attributed to compounds of similar chemical or biological composition to bevacizumab (including products derived from Chinese hamster ovary cells), doxorubicin, or dexrazoxane
* No HIV-positive patients receiving combination antiretroviral therapy
* No ongoing or active infection
* No psychiatric illness or social situations that would preclude study entry
* No other uncontrolled concurrent illness
* No serious, non-healing wound ulcer or bone fracture
* No significant traumatic injury within the past 3 weeks
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Chemotherapy
* At least 4 weeks since prior immunotherapy and recovered
* No other concurrent immunotherapy

Chemotherapy

* No prior doxorubicin or any other anthracyclines
* No more than 1 prior chemotherapy regimen

  * The following are not considered prior chemotherapy:

    * Immunotherapy, including cytokines
    * Peroxisome-proliferator-activated receptor gamma agonists or thalidomide
* At least 4 weeks since prior chemotherapy (6 weeks for carmustine or mitomycin) and recovered
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* At least 4 weeks since prior radiotherapy and recovered
* No concurrent radiotherapy

Surgery

* At least 3 weeks since prior major surgical procedure or open biopsy
* At least 1 week since prior needle biopsy

Other

* No other concurrent investigational agents
* No concurrent full-dose anticoagulants (except to maintain patency of preexisting, permanent indwelling IV catheters) or thrombolytic agent

  * Concurrent warfarin allowed if INR less than 1.5
* No concurrent chronic daily aspirin (more than 325 mg/day) or nonsteroidal anti -inflammatory medications known to inhibit platelet function
* No other concurrent investigational or commercial agents or therapies for this malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Maki, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Result] D'Adamo DR, Anderson SE, Albritton K, Yamada J, Riedel E, Scheu K, Schwartz GK, Chen H, Maki RG. Phase II study of doxorubicin and bevacizumab for patients with metastatic soft-tissue sarcomas. J Clin Oncol. 2005 Oct 1;23(28):7135-42. doi: 10.1200/JCO.2005.16.139. PMID 16192597